CLINICAL TRIAL: NCT01526850
Title: Phase Ⅱ/Ⅲ Clinical Trial, Multicenter, Randomized, Controlled, for the Evaluation of Efficacy and Safety of Therapy With Allogenic Mesenchymal Stem Cells in Patients With Chronic Graft Versus Host Disease
Brief Title: Efficacy and Safety Study of Allogenic Mesenchymal Stem Cells for Patients With Chronic Graft Versus Host Disease
Acronym: MSCsTcGVHD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Zhejiang University (Other); Chinese PLA General Hospital (Other); 307 Hospital of PLA (Other); Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Robert Chunhua Zhao, MD, PhD, MD, PhD，Professor of medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D07050701350701
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Cyclosporine; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allogenic mesenchymal stem cells (MSCs) (Experimental): patients who have developed an extensive chronic graft versus host disease (with skin and/or liver damage) after HSCs transplantation and do not respond to standard first-line regimen including cyclophosphamide and prednisolone.
  Interventions: Biological: Biological: mesenchymal stem cell
- Control group (Active Comparator): patients who have developed an extensive chronic graft versus host disease (with skin and/or liver damage) after HSCs transplantation and do not respond to standard first-line regimen including cyclophosphamide and prednisolone.
  Interventions: Drug: Cyclosporine and Glucocorticoid

INTERVENTIONS:
Biological: Biological: mesenchymal stem cell — Mesenchymal stem cells, 1-2×107, bone marrow injection, once a week for the first four weeks; whether to continue after four weeks depends on patients' symptoms.
  Other Names: Regenerative medicine: MSCs
  Arms: allogenic mesenchymal stem cells (MSCs)
Drug: Cyclosporine and Glucocorticoid — Calmodulin inhibitors such as cyclosporine, combined with Glucocorticoid 0.5-1mg/kg/d ,to the end of the study.
  Other Names: Calmodulin inhibitors combined with Glucocorticoid
  Arms: Control group

SUMMARY:
The primary purpose of the study is to evaluate the safety and efficacy of mesenchymal stem cells (MSC) for the treatment of patients who have developed an extensive chronic graft versus host disease (with skin and/or liver damage) after HSCs transplantation and do not respond to first-line therapy.

The secondary purpose of the study is to evaluate the effect of mesenchymal stem cells (MSC) on one-year survival rate, long-term survival rate, life quality and recurrence of patients who have developed an extensive chronic graft versus host disease (with skin and/or liver damage) after HSCs transplantation and do not respond to hormone treatment.

DETAILED DESCRIPTION:
Chronic Graft-versus-host disease (GVHD)， with the incidence of 30%-60%, is a serious late complication of allogeneic hematopoietic stem cell transplantation (HSCT) and is the major cause of death in the late stage of transplantation. According to targeted organs, cGVHD is divided into two types, limited cGVHD and extensive cGVHD. Extensive cGVHD needs systemic immunosuppressant treatment. However, currently standard first-line regimen including cyclophosphamide and prednisolone is only effective for some patients. Novel treatment is urgently needed. Our previous study has shown that mesenchymal stem cells (MSCs) are effective for cGVHD patients with multiple skin damage. To further explore the therapeutic effect of MSCs for extensive cGVHD, we plan to conduct a multi-center clinical trial. Patients who developed an extensive cGVHD (with skin and/or liver damage) after HSCs transplantation and do not respond to first-line therapy are enrolled. They will be randomly divided into two groups which will receive MSCs and routine second-line drugs respectively. We will evaluate the efficacy and safety of MSCs for extensive cGVHD by comparison of symptom improvement, survival rate, recurrence as well as side effects in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Extensive cGVHD with skin and/or liver damage developed after allogeneic hematopoietic stem cell transplantation
* cGVHD that do not response to conventional immunosuppressant treatment for two months
* KPS>= 30
* informed consent from the patient

Exclusion Criteria:

* Extensive cGVHD without skin or liver damage
* With other acute severe complications
* In pregnancy or lactation
* Disease relapses
* With non-hematological malignancy
* Have a history of mental disorder, drug or alcohol abuse over the past five years
* Allergic
* Participate in other clinical trial within three months before the start of this trial
* With bone marrow fibrosis
* Have undergone hematopoietic stem cell transplantation to treat solid tumor

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The total Response rate defined as patients with complete and partial response | 1 year after MSCs administration.

SECONDARY OUTCOMES:
one-year survival rate | 1 year after MSCs administration
disease relapse | 2 years after MSCs administration
quality of life | 2 years after MSCs administration

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University; Chunhua Zhao, MD,PHD, Principal Investigator — Peking Union Medical College
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Sun Z, Han Q, Zhu Y, Li Z, Chen B, Liao L, Bian C, Li J, Shao C, Zhao RC. NANOG has a role in mesenchymal stem cells' immunomodulatory effect. Stem Cells Dev. 2011 Sep;20(9):1521-8. doi: 10.1089/scd.2010.0366. Epub 2011 Feb 26. PMID 21235326
- [Background] Shi D, Liao L, Zhang B, Liu R, Dou X, Li J, Zhu X, Yu L, Chen D, Zhao RC. Human adipose tissue-derived mesenchymal stem cells facilitate the immunosuppressive effect of cyclosporin A on T lymphocytes through Jagged-1-mediated inhibition of NF-kappaB signaling. Exp Hematol. 2011 Feb;39(2):214-224.e1. doi: 10.1016/j.exphem.2010.10.009. Epub 2010 Nov 13. PMID 21078360
- [Background] Liu K, Chen Y, Zeng Y, Xu L, Liu D, Chen H, Zhang X, Han W, Wang Y, Zhao T, Wang J, Wang J, Han Q, Zhao C, Huang X. Coinfusion of mesenchymal stromal cells facilitates platelet recovery without increasing leukemia recurrence in haploidentical hematopoietic stem cell transplantation: a randomized, controlled clinical study. Stem Cells Dev. 2011 Oct;20(10):1679-85. doi: 10.1089/scd.2010.0447. Epub 2011 Feb 5. PMID 21142788
- [Background] Wu Y, Zhao RC, Tredget EE. Concise review: bone marrow-derived stem/progenitor cells in cutaneous repair and regeneration. Stem Cells. 2010 May;28(5):905-15. doi: 10.1002/stem.420. PMID 20474078
- [Background] Zhou H, Guo M, Bian C, Sun Z, Yang Z, Zeng Y, Ai H, Zhao RC. Efficacy of bone marrow-derived mesenchymal stem cells in the treatment of sclerodermatous chronic graft-versus-host disease: clinical report. Biol Blood Marrow Transplant. 2010 Mar;16(3):403-12. doi: 10.1016/j.bbmt.2009.11.006. Epub 2009 Nov 17. PMID 19925878
- [Background] Guo M, Sun Z, Sun QY, Han Q, Yu CL, Wang DH, Qiao JH, Chen B, Sun WJ, Hu KX, Liu GX, Liu B, Zhao RC, Ai H. A modified haploidentical nonmyeloablative transplantation without T cell depletion for high-risk acute leukemia: successful engraftment and mild GVHD. Biol Blood Marrow Transplant. 2009 Aug;15(8):930-7. doi: 10.1016/j.bbmt.2009.04.006. PMID 19589482
- [Background] Zhu Y, Sun Z, Han Q, Liao L, Wang J, Bian C, Li J, Yan X, Liu Y, Shao C, Zhao RC. Human mesenchymal stem cells inhibit cancer cell proliferation by secreting DKK-1. Leukemia. 2009 May;23(5):925-33. doi: 10.1038/leu.2008.384. Epub 2009 Jan 15. PMID 19148141
- [Background] Zhang B, Liu R, Shi D, Liu X, Chen Y, Dou X, Zhu X, Lu C, Liang W, Liao L, Zenke M, Zhao RC. Mesenchymal stem cells induce mature dendritic cells into a novel Jagged-2-dependent regulatory dendritic cell population. Blood. 2009 Jan 1;113(1):46-57. doi: 10.1182/blood-2008-04-154138. Epub 2008 Oct 2. PMID 18832657
- [Background] Liao L, Zhao RC. An overview of stem cell-based clinical trials in China. Stem Cells Dev. 2008 Aug;17(4):613-8. doi: 10.1089/scd.2008.0183. PMID 18673001
- [Background] Ren G, Zhang L, Zhao X, Xu G, Zhang Y, Roberts AI, Zhao RC, Shi Y. Mesenchymal stem cell-mediated immunosuppression occurs via concerted action of chemokines and nitric oxide. Cell Stem Cell. 2008 Feb 7;2(2):141-50. doi: 10.1016/j.stem.2007.11.014. PMID 18371435
- [Background] Chen L, Zhang W, Yue H, Han Q, Chen B, Shi M, Li J, Li B, You S, Shi Y, Zhao RC. Effects of human mesenchymal stem cells on the differentiation of dendritic cells from CD34+ cells. Stem Cells Dev. 2007 Oct;16(5):719-31. doi: 10.1089/scd.2007.0065. PMID 17999594
- [Background] Deng W, Han Q, Liao L, You S, Deng H, Zhao RC. Effects of allogeneic bone marrow-derived mesenchymal stem cells on T and B lymphocytes from BXSB mice. DNA Cell Biol. 2005 Jul;24(7):458-63. doi: 10.1089/dna.2005.24.458. PMID 16008514
- [Background] Deng W, Han Q, Liao L, Li C, Ge W, Zhao Z, You S, Deng H, Zhao RC. Allogeneic bone marrow-derived flk-1+Sca-1- mesenchymal stem cells leads to stable mixed chimerism and donor-specific tolerance. Exp Hematol. 2004 Sep;32(9):861-7. doi: 10.1016/j.exphem.2004.06.009. PMID 15345288
- [Background] Zhang W, Ge W, Li C, You S, Liao L, Han Q, Deng W, Zhao RC. Effects of mesenchymal stem cells on differentiation, maturation, and function of human monocyte-derived dendritic cells. Stem Cells Dev. 2004 Jun;13(3):263-71. doi: 10.1089/154732804323099190. PMID 15186722